CLINICAL TRIAL: NCT07335887
Title: An Optimized Treatment for Patients With Primary Systemic Light Chain Amyloidosis
Brief Title: Sonrotoclax Plus Dexamethasone With or Without Daratumumab Regimen in Patients With t(11;14) Primary AL Amyloidosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, chief physician, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025PHD030-002
Record Dates: First submitted 2025-12-14; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: AL Amyloidosis (AL); t(11;14) Positive
Keywords: sonrotoclax; AL amyloidosis; t(11;14); BCL-2i
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — daratumumab; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sond±D (Experimental): Cohort A: sonrotoclax combined with daratumumab and dexamethasone in t(11;14) AL amyloidosis, newly diagnosed or previously untreated with anti-CD38 mAb therapy.
  Cohort B: sonrotoclax combined with daratumumab and dexamethasone in t(11;14) AL patients insensitive to or relapsed after anti-CD38 mAb therapy
  Interventions: Drug: sonrotoclax; Drug: Daratumumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: sonrotoclax — t(11;14) AL amyloidosis Newly diagnosed or previously untreated with anti-CD38 mAb therapy
  Induction therapy (C1-4) Sonrotoclax once daily ( dose depends on the 3+3 study design during safety run-in period in C1)
  Consolidation therapy (C5-12) Sonrotoclax once daily (same as the target dose in induction therapy)
  t(11;14) AL patients insensitive to or relapsed after anti-CD38 mAb therapy
  Induction therapy (C1-4) Sonrotoclax once daily (dose depends on the 3+3 study design during safety run-in period in C1)
  Consolidation therapy (C5-12) Sonrotoclax once daily (same as the target dose in induction therapy)
  Other Names: BGB-11417
Drug: Daratumumab — t(11;14) AL patients insensitive to or relapsed after anti-CD38 mAb therapy
  Daratumumab (16 mg/kg intravenously or 1800 mg subcutaneously, once weekly C1-2; every two weeks C3-6; every month C7-12)
Drug: Dexamethasone — Dexamethasone (40 mg, once weekly) for 12 cycles. The dose was halved for patients 75 years of age or older, and in patients who were intolerant of dexamethasone, as judged by the investigators.

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of Sonrotoclax combined Regimen in patients with t(11;14) AL amyloidosis. Participants will receive the Sonrotoclax Plus Dexamethasone regimen with or without Daratumumab for 12 cycles. The Hematologic Response, Organ Response, Survival, and Safety will be evaluated.

DETAILED DESCRIPTION:
Treatment options for AL amyloidosis are limited. Before the approval of daratumumab, newly diagnosed light-chain amyloidosis was often managed with anti-myeloma regimens such as bortezomib. For patients with relapsed/refractory (R/R) disease, there is currently a lack of standard treatment options both domestically and internationally. Guidelines recommend enrollment in clinical trials or the use of regimens containing previously unexposed agents, such as bortezomib or daratumumab.

Based on preliminary data of BCL-2 inhibitors in t(11;14) amyloidosis, this study aims to explore the efficacy and safety of sonrotoclax and dexamethasone with or without Daratumumab. Newly diagnosed patients with t（11;14）will receive the combination of sonrotoclax, daratumumab, and dexamethasone. t(11;14) Patients with relapsed/refractory AL amyloidosis (RRAL) will be treated with sonrotoclax plus dexamethasone. For transplant-eligible patients, stem cell collection is permitted during the induction phase of therapy. The timing of ASCT may be assessed after the primary endpoint evaluation (completion of 4 treatment cycles) and determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria for Primary Systemic Light Chain Amyloidosis (according to the Systemic Light Chain Amyloidosis Diagnosis and Treatment Guidelines (2021 Revision)).
2. Age ≥ 18 years.
3. Confirmed FISH test result of t(11;14) positive by each center or a third-party laboratory, or a prior FISH test report indicating t(11;14) positivity
4. ECOG Performance Status score of 0-2.
5. Presence of measurable disease, defined by at least one of the following criteria:

   1. Serum M-protein ≥ 0.5 g/dL
   2. Serum free light chain (FLC) level ≥ 40 mg/L with an abnormal kappa/lambda ratio.
6. Adequate organ function, defined as:

   1. Hemoglobin (HGB) > 80 g/L
   2. Platelet count > 50 × 10⁹/L
   3. Absolute neutrophil count (ANC) > 1.0 × 10⁹/L
   4. Total bilirubin ≤ 2.0 × ULN; AST and ALT ≤ 3.0 × ULN
   5. Creatinine clearance (CrCl) ≥ 30 mL/min
   6. Oxygen saturation ≥ 90%
7. Life expectancy greater than 6 months.
8. Patient understands and voluntarily signs an informed consent form (ICF).
9. Cohort Assignment:

   * Cohort A: Includes patients who are newly diagnosed or have not been previously exposed to anti-CD38 monoclonal antibody therapy.
   * Cohort B: Includes patients who are insensitive to or have relapsed after anti-CD38 monoclonal antibody therapy.Insensitivity to anti-CD38 monoclonal antibody therapy is defined as failure to achieve at least a Partial Response (PR) after 1 cycle, or failure to achieve at least a Very Good Partial Response (VGPR) after 3 cycles of an anti-CD38-containing regimen.

Exclusion Criteria:

1. Meets the diagnostic criteria for active multiple myeloma or active lymphoplasmacytic lymphoma
2. Presence of other malignancies at an advanced stage with systemic metastases.
3. IgM-type AL amyloidosis.
4. Prior treatment with a BCL-2 inhibitor (BCL-2i).
5. Presence of any of the following severe cardiovascular diseases

   1. Mayo 2004 stage IIIb: NT-proBNP >8500 ng/L.
   2. NYHA class IIIb-IV
   3. Left ventricular ejection fraction (LVEF) <40%.
   4. QT interval corrected by Fridericia's formula (QTcF) >480 ms
   5. Investigator assessment that heart failure is due to ischemic heart disease (e.g., prior history of myocardial infarction with elevated cardiac enzymes and ECG changes) or uncorrected valvular disease, rather than primarily caused by AL amyloidosis.
   6. Hospitalization for unstable angina or myocardial infarction within 6 months prior to the first dose, or cardiac interventional therapy or coronary artery bypass grafting within 6 months.
   7. For patients with congestive heart failure, hospitalization for cardiovascular disease within 4 weeks prior to Cycle 1 Day 1.
   8. History of sustained ventricular tachycardia or aborted ventricular fibrillation, or history of atrioventricular node or sinus node dysfunction requiring a pacemaker/implantable cardioverter-defibrillator (ICD) but not implanted.
6. Severe or persistent infection that is not effectively controlled. (Acute infection requiring antibacterial, antifungal, or antiviral therapy that has not resolved within 14 days prior to dosing).
7. Positive status for human immunodeficiency virus (HIV) antibody (HIVAb).
8. Serological status reflecting active viral hepatitis B (HBV) or hepatitis C (HCV) infection, as follows:

   1. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Patients who are positive for HBcAb but negative for HBsAg are eligible if HBV DNA is undetectable and they are willing to undergo monthly monitoring for HBV reactivation.
   2. Positive for hepatitis C virus (HCV) antibody. Patients who are positive for HCV antibody are eligible if HCV RNA is undetectable.
9. Patients receiving renal replacement therapy.
10. Patients with known hypersensitivity to any component of the investigational regimen.
11. Any condition that, in the investigator's judgment, would increase the risk to the subject or affect the study results.
12. Patients with AL amyloidosis currently participating in other investigational drug clinical studies.
13. Patients who are pregnant, breastfeeding, or planning to become pregnant during the study participation.
14. Patients who are receiving any moderate or strong CYP3A4 inhibitors (within ≤7 days or 5 half-lives, whichever is shorter) or strong CYP3A4 inducers (within ≤14 days or 5 half-lives, whichever is shorter) prior to the first dose of the study drug; or patients who require continuous treatment with moderate or strong CYP3A inhibitors or strong CYP3A inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Best hematological ≥VGPR rate within four cycles of therapy | At the end of Cycle 4 (each cycle is 28 days)
  Defined as the proportion of patients achieving VGPR, or CR within four cycles of therapy

SECONDARY OUTCOMES:
Hematological ORR after four cycles of therapy | At the end of Cycle 4 (each cycle is 28 days)
  Defined as the proportion of patients achieving PR,VGPR, or CR at the end of four cycles of therapy
Hematological CR rate at the end of four cycles of therapy | at the end of 4 cycles of therapy (each cycle is 28 days)
  Defined as the proportion of patients achieving CR at the end of four cycles of therapy
Cardiac response rate at the end of 6 cycles of treatment | At the end of Cycle 6 (each cycle is 28 days)
  Defined as the proportion of patients achieving Cardiac response at the end of 6 cycles of therapy
Hepatic response rate at the end of 6 cycles of treatment | At the end of Cycle 6 (each cycle is 28 days)
  Defined as the proportion of patients achieving Hepatic response at the end of 6 cycles of therapy
Renal response rate at the end of 6 cycles of treatment | At the end of 6 cycles of treatment (each cycle is 28 days)
  Defined as the proportion of patients achieving Hepatic response at the end of 6 cycles of therapy
1-year MOD-PFS rate | 1 year
  Defined as the proportion of patients in the safety analysis set who have not experienced a MOD-PFS event within 1 year after treatment. MOD-PFS is defined as the time from treatment initiation to the occurrence of any of the following events (whichever comes first): end-stage heart disease (requiring heart transplantation, left ventricular assist device, or intra-aortic balloon pump), end-stage renal disease (requiring dialysis or renal transplantation), hematological progression, or death
1-year PFS rate | 1 year
  Defined as the proportion of patients in the safety analysis set who are alive and free from hematological progression at 1 year after treatment. PFS is defined as the time from treatment initiation to hematological progression or death (whichever occurs first)
1-year OS rate | 1 year
  Defined as the proportion of patients in the safety analysis set who are alive at 1 year after treatment
Time to Response (TTR) | 1 year
  Defined as the time from treatment initiation to the first hematological efficacy assessment achieving PR.
Time to VGPR | 1 year
  Defined as the time from treatment initiation to the first hematological efficacy assessment achieving VGPR
Time to Cardiac Response | 1 year
  Defined as the time from treatment initiation to the first cardiac efficacy assessment achieving response.
Time to Renal Response | 1 year
  Defined as the time from treatment initiation to the first renal efficacy assessment achieving response
Time to Hepatic Response | 1 year
  Defined as the time from treatment initiation to the first hepatic efficacy assessment achieving response.
Adverse Events (AEs), Serious Adverse Events (SAEs), and laboratory abnormalities | 1 year
  the proportion of patients with Adverse Events (AEs), Serious Adverse Events (SAEs), and laboratory abnormalities after therapy
Correlation analysis between different MRD satus groups and MOD-PFS, PFS and OS | 1 year
  Correlation analysis between different MRD satus groups and 1-year MOD-PFS, 1-year PFS and 1-year OS

OTHER OUTCOMES:
MRD negativity rate in patients achieving hematological CR | 1 year
  Defined as the MRD negativity rate in patients achieving hematological CR
MRD negativity rate | At the end of Cycle 9-12 (each cycle is 28 days)
  Defined as the proportion of patients achieving MRD negativity